CLINICAL TRIAL: NCT06645145
Title: Language Experience and Language Learning
Brief Title: Language Learning and Language Experience
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Montclair State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-FY24-25-3948
Record Dates: First submitted 2024-10-03; First posted 2024-10-16 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Typically Developing Children Ages 3 to 6
Keywords: verb learning; orthographic facilitation; typical development

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Verb learning with only visual and auditory support (No Intervention): This is "gold standard" learning scenario for young children.
- Verb learning with auditory, visual, and text support (Experimental): Participants receive the added support of text to determine if this additional support helps them learn novel words with higher accuracy.
  Interventions: Behavioral: Orthographic facilitation

INTERVENTIONS:
Behavioral: Orthographic facilitation — Half of participants will receive orthographic support (text support) while learning new verbs. The investigators will compare learning with and without text support to determine if this aids verb learning.
  Arms: Verb learning with auditory, visual, and text support

SUMMARY:
The goal of this clinical trial is to learn if text can support children in learning new verbs in healthy children ages three through six. The main questions it aims to answer are:

Does text support help children learn new verbs? Does a child's relative benefit from text support vary according to their literacy skills?

Participants will

* Watch videos of actions and hear novel words
* Name alphabet sounds to determine their literacy skills

ELIGIBILITY:
Inclusion Criteria:

* Primarily exposed to English
* Typical development
* Hearing and vision within normal limits or corrected to be so

Ages: 36 Months to 84 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 170 (Actual)
Dates: Start 2024-10-31 (Actual); Primary Completion 2025-08-30 (Actual); Study Completion 2025-08-30 (Actual)

PRIMARY OUTCOMES:
Accuracy | 15 minutes
  The investigators will measure accuracy in an identification task with a pointing response.

SECONDARY OUTCOMES:
Literacy as a Mediator | 15 minutes
  The investigators will compare orthographic facilitation across literacy measures to determine if/how literacy mediates how much of an effect text support offers.

CONTACTS AND LOCATIONS:
Overall Officials: Grace Clark, PhD, Principal Investigator — Montclair State University
Locations (1):
- Online Asynchronous, Bloomfield, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data will be sent upon request.
Supporting Information: Study Protocol, CSR, Analytic Code